CLINICAL TRIAL: NCT02461433
Title: The SAVIOR Trial: Surgical Application of Vac Dressings In Obese Patients to Reduce Wound Complications
Brief Title: Surgical Application of Vac Dressings In Obese Patients to Reduce Wound Complications
Acronym: SAVIOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor pulled funding
Sponsor: Johns Hopkins University (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00030337
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Wound Infection, Surgical; Obesity; Postoperative Complications
Keywords: Obesity; Obese; surgical site infection; closed incisions; negative pressure therapy
MeSH Terms: conditions — Surgical Wound Infection; Obesity; Postoperative Complications

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Prevena (Experimental): After surgery this group will receive the Prevena device (negative pressure wound therapy).
  Interventions: Device: Prevena
- Standard dressing (Active Comparator): After surgery this group will receive standard of care dressings on their surgical wound.
  Interventions: Device: Standard Dressing

INTERVENTIONS:
Device: Prevena — Prevena Incision Management system
  Arms: Prevena
Device: Standard Dressing — This involves standard of care dressing including but not limited to gauze.
  Arms: Standard dressing

SUMMARY:
The purpose of this study is to determine whether application of an incisional wound Prevena trademark (TM) dressing (applies negative pressure to wounds) in the obese (BMI ≥30) surgical patient will reduce surgical site infections (SSI) when compared to the standard of care dressing.

DETAILED DESCRIPTION:
In an attempt to decrease wound infection incidence and improve healing time of open surgical wounds, vacuum assisted closure (VAC) was developed. This innovative technique provided contained controlled wound irrigation without bacterial aerosolization. A newer customizable subset of the Prevena incision Management System TM called Prevena Peel and Place TM has been released a few months ago. The new model can be cut to specific wound sizes and has a connector that can be attached to the already widely available VAC machines. The versatility and the comparability to older models of Prevena Peel and Place TM have not been tested to this date.

The investigators believe that a randomized clinical trial evaluating the use of the Prevena Incision Management System TM for homecare and the use of Prevena Peel and Place TM for inpatients in special populations is warranted. Obese patients (BMI≥30) undergoing open surgery will have decreased surgical site infection rates, improved healing time, better quality of life (QOL) and lower readmission rates with use of Prevena in the post-operative management of surgical incisions.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been informed of the nature of the study, and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) / Medical Ethics Committee (MEC) of the respective clinical site.
* Patient meets the criteria for and is undergoing open surgery at Johns Hopkins Medical Institutes.
* Patient with BMI≥ 30 at the time of surgery
* Patient agrees to return for all required clinical follow up for the study.

Exclusion Criteria:

* Known allergic reaction to acrylic adhesives or silver.
* Known history of intolerance to any component of Prevena Incision Management System TM.
* Very fragile skin around incision site.
* Bleeding disorder or refuses blood transfusion.
* Malignancy or other condition limiting life expectancy to <5 years.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley Steele, MD, PHD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutes, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevena | Standard Dressing
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevena | Standard Dressing | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 34 [34 to 34] | 45 [45 to 45] | 39.5 [34 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants] — Location of where the participant was enrolled.
  Participants
    United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Surgical Site Infection According to National Healthcare Safety Network - Center for Disease Control Guidelines
Description: The incidence of postoperative surgical site infection (according to National Healthcare Safety Network - Center for Disease Control guidelines) in open surgery
Time Frame: Up to 7 days postop
Measure: Number; unit: Surgical Site infections
Arm/Group | Prevena | Standard Dressing
Number analyzed (Participants) | 1 | 1
Surgical Site infections | 0 | 0

2. Secondary Outcome: Other Wound Complications (Aggregate)
Description: Dehiscence, seroma and hematoma. Reported as number of aggregate events.
Time Frame: Up to 14 days postop
Measure: Number; unit: aggregate wound complication events
Arm/Group | Prevena | Standard Dressing
Number analyzed (Participants) | 1 | 1
aggregate wound complication events | 0 | 0

3. Secondary Outcome: Skin Bacterial Count as Assessed by Microbacterial Count
Description: Skin bacterial count after removal of either Prevena or standard dressing. A micro-bacterial swap will be performed and sent to the microbiology lab for assessing bacterial count
Time Frame: Up to 7 days postop
Population: The samples were not sent to the lab
Arm/Group | Prevena | Standard Dressing
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Physical Function as Assessed by Short Form Survey (SF) 36
Description: The SF -36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability
Time Frame: Up to 14 days postop
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Prevena | Standard Dressing
Number analyzed (Participants) | 1 | 1
units on a scale | 100 [100 to 100] | 85 [85 to 85]

5. Secondary Outcome: Readmissions
Description: Readmission events for the patients.
Time Frame: Up to 30 days postop
Measure: Number; unit: readmission events
Arm/Group | Prevena | Standard Dressing
Number analyzed (Participants) | 1 | 1
readmission events | 0 | 0

6. Secondary Outcome: Role Limitations Due to Physical Health as Assessed by Short Form Survey (SF) 36
Description: as for outcome 4
Time Frame: Up to 14 days postop
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Prevena | Standard Dressing
Number analyzed (Participants) | 1 | 1
units on a scale | 100 [100 to 100] | 100 [100 to 100]

7. Secondary Outcome: Social Functioning as Assessed by Short Form Survey (SF) 36
Description: as for outcome 4
Time Frame: Up to 14 days postop
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Prevena | Standard Dressing
Number analyzed (Participants) | 1 | 1
units on a scale | 100 [100 to 100] | 100 [100 to 100]

8. Secondary Outcome: Energy / Fatigue as Assessed by Short Form Survey (SF) 36
Description: The SF -36 has eight scaled scores; the scores are weighted sums of the questions in each section. Energy and fatigue are aggregated in this section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability
Time Frame: Up to 14 days postop
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Prevena | Standard Dressing
Number analyzed (Participants) | 1 | 1
units on a scale | 50 [50 to 50] | 75 [75 to 75]

9. Secondary Outcome: Emotional Well Being as Assessed by Short Form Survey (SF) 36
Description: as for outcome 4
Time Frame: Up to 14 days postop
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Prevena | Standard Dressing
Number analyzed (Participants) | 1 | 1
units on a scale | 60 [60 to 60] | 60 [60 to 60]

10. Secondary Outcome: Pain as Assessed by Short Form Survey (SF) 36
Description: as for outcome 4
Time Frame: Up to 14 days postop
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Prevena | Standard Dressing
Number analyzed (Participants) | 1 | 1
units on a scale | 100 [100 to 100] | 100 [100 to 100]

11. Secondary Outcome: General Health as Assessed by Short Form Survey (SF) 36
Description: as for outcome 4
Time Frame: Up to 14 days postop
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Prevena | Standard Dressing
Number analyzed (Participants) | 1 | 1
units on a scale | 100 [100 to 100] | 65 [65 to 65]

ADVERSE EVENTS:
Time Frame: From consent to end of study (30 days)
Description: Used a checklist to inquire about would feeling, and systemic effects
Arm/Group | Prevena | Standard Dressing
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT02461433/Prot_SAP_000.pdf